CLINICAL TRIAL: NCT04537962
Title: Avaliação da Carga do vírus SARS-CoV-2 na Cavidade Oral e na Saliva após desinfecção Com soluções Antimicrobianas Orais e dentifrícios.
Brief Title: Salivary SARS-CoV-2 Load of Covid-19 Patients After Oral Antimicrobial Solutions and Dentifrices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4172-20
Record Dates: First submitted 2020-07-14; First posted 2020-09-03 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2020-07

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Toothpastes; fluorophosphate; Sodium Fluoride; Zinc; Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Colgate Periogard and Peroxyl® (Placebo Comparator): Patients hospitalized in the ICU with orotracheal intubation or negative pressure room - will undergo antisepsia of the oral mucosa with 1.5% hydrogen peroxide solution, following by a 0.12% non-alcoholic chlorhexidine solution
  Interventions: Other: Colgate Periogard® mouthwash; Other: Colgate Peroxyl® mouthwash
- Colgate Periogard® (Placebo Comparator): Patients hospitalized in the ICU with orotracheal intubation or negative pressure room - will undergo antisepsia of the oral mucosa with 0.12% non-alcoholic chlorhexidine solution;
  Interventions: Other: Colgate Periogard® mouthwash
- Colgate Peroxyl® (Placebo Comparator): Patients hospitalized in negative pressure rooms - will undergo antisepsia of the oral mucosa with 1.5% hydrogen peroxide solution
  Interventions: Other: Colgate Peroxyl® mouthwash
- Colgate Total 12® (Placebo Comparator): Patients hospitalized in negative pressure rooms - will undergo antisepsia of the oral mucosa with 0.075% cetylpyridinium chloride associated with 0.28% zinc lactate
  Interventions: Other: Colgate Total® Mouthwash
- Toothpaste with sodium monofluorophosphate (Active Comparator): Patients hospitalized in negative pressure rooms - will undergo brushing with dentifrice containing only 1.1% fluoride, water, glycerin, cellulose, sodium lauryl sulfate, and sodium bicarbonate
  Interventions: Other: Toothpaste with sodium monofluorophosphate
- Toothpaste with sodium fluoride and zinc (Active Comparator): Patients hospitalized in negative pressure rooms - will undergo brushing with dentifrice containing 0.32% fluoride, 0.96% zinc, arginine, poloxamer, glycerin, water, hydrated silica, sodium lauryl sulfate, and sodium saccharin
  Interventions: Other: Toothpaste with sodium fluoride and zinc
- Toothpaste with tin fluoride (Active Comparator): Patients hospitalized in negative pressure rooms - will undergo brushing with dentifrice containing 0.454% stannous fluoride, water, sorbitol, hydrated silica, glycerin, tetrasodium pyrophosphate, microcrystalline cellulose, and xanthan gum
  Interventions: Other: Toothpaste with tin fluoride

INTERVENTIONS:
Other: Colgate Periogard® mouthwash — Patients will be submitted to antisepsia of the oral mucosa with Colgate Periogard® mouthwash
  Arms: Colgate Periogard and Peroxyl®; Colgate Periogard®
Other: Colgate Peroxyl® mouthwash — Patients will be submitted to antisepsia of the oral mucosa with Colgate Peroxyl® mouthwash
  Arms: Colgate Periogard and Peroxyl®; Colgate Peroxyl®
Other: Colgate Total® Mouthwash — Patients will be submitted to antisepsia of the oral mucosa with Colgate Total® Mouthwash
  Arms: Colgate Total 12®
Other: Toothpaste with sodium monofluorophosphate — Patients will be submitted to brushing with toothpaste with sodium monofluorophosphate
  Arms: Toothpaste with sodium monofluorophosphate
Other: Toothpaste with sodium fluoride and zinc — Patients will be submitted to brushing with toothpaste with sodium fluoride and zinc
  Arms: Toothpaste with sodium fluoride and zinc
Other: Toothpaste with tin fluoride — Patients will be submitted to brushing with toothpaste with tin fluoride
  Arms: Toothpaste with tin fluoride

SUMMARY:
The aim of this study is to analyze if the use of oral antimicrobial solutions and dentifricies are able to reduce the SARS-CoV-2 load in the saliva and oral mucosa. It will be allocated hospitalized patients positive for SARS-CoV-2 (confirmed by RT-PCR of nasopharynx swab tests) and with signs and symptoms of COVID-19. These patients will be divided into two groups: patients enrolled in negative pressure rooms (NPR), and patients enrolled in intensive care units (ICU) with orotracheal intubation. These two groups will receive interventions with oral antimicrobial solutions or dentifrices, containing different compounds. Saliva and oral mucosa swabs will be collected before the intervention, immediately after the intervention, and after 30min and 1h. The primary outcome is to verify if these products can reduce the SARS-CoV-2 load in the saliva and oral mucosa at these time periods, detected by the measurement of the viral load and the fold-reduction.

DETAILED DESCRIPTION:
Each group of patients will receive specific interventions, as follows:

NPR group (n=60) - three interventions with different mouthwashes solutions (12 patients in each intervention): 1) 0.12% chlorhexidine solution (Colgate Periogard®); 2) mouthwash with 1.5% hydrogen peroxide solution (Colgate Peroxyl®); 3) mouthwash with 0.075% cetylpyridinium chloride solution (Colgate Total 12®); 4) 1.5% hydrogen peroxide solution plus 0.12% chlorhexidine solution (Colgate Peroxyl® followed by Colgate Periogard®).

The interventions will be compared with a Placebo, which will be a mouthwash with distilled water (n=12).

NPR group (n=90) - three interventions with different dentifrices (30 patients in each intervention): 1) dentifrice containing only 1.1% fluoride, water, glycerin, cellulose, sodium lauryl sulfate, and sodium bicarbonate; 2) dentifrice containing 0.32% fluoride, 0.96% zinc, arginine, poloxamer, glycerin, water, hydrated silica, sodium lauryl sulfate, and sodium saccharin 3) dentifrice containing 0.454% stannous fluoride, water, sorbitol, hydrated silica, glycerin, tetrasodium pyrophosphate, microcrystalline cellulose, and xanthan gum .

The interventions will be compared to each other. ICU group (n=52)- two interventions with different oral antimicrobial solutions (26 patients in each intervention): 1) 0.12% chlorhexidine solution (Colgate Periogard®); 2) 1.5% hydrogen peroxide solution plus 0.12% chlorhexidine solution (Colgate Peroxyl® followed by Colgate Periogard®).

The interventions will be compared to each other.

ELIGIBILITY:
Inclusion Criteria:

* Patients positive for SARS-CoV-2 using the RT-PCR method and requiring oral hygiene care and other preventive and therapeutic dental procedures.

Exclusion Criteria:

* Pediatric patients, negative for SARS-CoV-2 by the RT-PCR method, exhibiting oral ulcerations and other erosive lesions in the oral mucosa that contraindicate the use of hydrogen peroxide, chlorhexidine and cetylpyridinium, patients who present bleeding in the oral cavity. that prevents the collection of samples, patients who report a history of allergy, irritations or other side effects derived from the use of these substances, who do not adhere to the oral care protocols or those in which it is not possible to perform these procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Reduction of SARS-CoV-2 load in the oral mucosa and saliva | 1 hour
  Reduction of SARS-CoV-2 load in the oral mucosa and saliva measured by viral fold-reduction and viral quantitation

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Correa, PhD, Study Director — University of Sao Paulo; Debora H Douek, PhD, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital israelita Albert Einstein, São Paulo, Brazil

REFERENCES:
- [Derived] Bezinelli LM, Correa L, Beyerstedt S, Franco ML, Rangel EB, Benitez CG, Hamerschlak N, Pinho JRR, Heller D, Eduardo FP. Reduction of SARS-CoV-2 viral load in saliva after rinsing with mouthwashes containing cetylpyridinium chloride: a randomized clinical study. PeerJ. 2023 Dec 18;11:e15080. doi: 10.7717/peerj.15080. eCollection 2023. PMID 38130922
- [Derived] Eduardo FP, Correa L, Mansur F, Benitez C, Hamerschlak N, Pinho JRR, Heller D, Bezinelli LM. Effectiveness of Toothpastes on SARS-CoV-2 Viral Load in Saliva. Int Dent J. 2022 Dec;72(6):825-831. doi: 10.1016/j.identj.2022.03.006. Epub 2022 Mar 23. PMID 35570015